CLINICAL TRIAL: NCT05582369
Title: Setting Expectations for Enjoyment of Physical Activity
Brief Title: Feel the Move: A Micro-Randomized Trial of a Text-Based Expectation-Setting Intervention to Increase Physical Activity
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Michigan (Other)
Responsible Party: Principal Investigator, Pedja Klasnja, Associate Professor, University of Michigan
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: HUM00190301
Record Dates: First submitted 2022-09-21; First posted 2022-10-17 (Actual); Last update posted 2024-06-25 (Actual); Status verified 2024-06

CONDITIONS: Physical Activity
MeSH Terms: conditions — Motor Activity

STUDY DESIGN:
Intervention Model Description: At each decision point-operationalized as the beginning of the time window during which a participant planned to exercise-each participant will be randomized to receive one of three intervention options: active intervention (text messages aimed to prime expectations of emotional rewards of exercise), a control message (a reminder that they will receive a study questionnaire later in the day), or no intervention.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Affective Rewards Messages (Experimental): Throughout the study, each week participants will be asked to plan two exercise sessions for the upcoming week, and will be asked to report on how they did with those plans at the end of the day when they planned to exercise. At the very beginning of the time window when they planned to exercise participants will be randomized with 40% probability to receive no message, 20% probability to receive a reminder to fill out the study questionnaire at the end of the day, and 40% probability to receive one of two types of affective rewards messages (active intervention). The two types are: 1) low-reflection messages written by participants at the beginning of the study, about the affective rewards of exercise they have previously experienced; and 2) high-reflection messages that prompt participants to reflect on the affective rewards of exercise and text back a response.
  Interventions: Behavioral: Affective Rewards Messages

INTERVENTIONS:
Behavioral: Affective Rewards Messages — Messages about the affective rewards of exercise

SUMMARY:
The aim of this research is to evaluate the impacts of an intervention that reminds people of the affective rewards of exercise on physical activity in adults of any activity level

DETAILED DESCRIPTION:
The Feel the Move study tests the effects of a lightweight text-message based intervention to increase physical activity and affective attitudes towards exercise. The intervention being investigated is text messages that prime expected affective rewards of exercise, sent in advance of a time window during which participants made plans to exercise. At the start of the study, participants will write sentences about feeling good after exercise (which will be used as part of the intervention) and complete baseline questionnaires about their feelings towards exercise. For the next nine weeks, participants will be asked to plan two exercise sessions a week, and will be given a questionnaire after the time window of their planned exercise sessions to assess how it went. At the onset of each time window for their planned exercise session, participants will be micro-randomized to receive one of the following intervention options: no-message; a text message reminding them to fill out the study questionnaires; or a message about the affective rewards of exercise. The messages about affective rewards will be a mix of sentences participants wrote themselves during the baseline assessment and reflective prompts from the research team. At the nine-week mark, participants will again complete the same questionnaires about their feelings towards exercise that they initially completed at baseline. Throughout the study, participants will share data about their activity, including steps and calories burned, with the research team. These data will be automatically collected by the HIPAA-compliant CareEvolution platform from participants' Apple Watches. After the nine weeks of the study participation, a random sample of study participants will be asked to participate in exit interviews to share more details about their experiences with the intervention.

The primary hypothesis is that participants will burn more calories during their planned exercise periods when they receive messages about the affective rewards of exercise vs. when they do not. Researchers will also conduct secondary analyses examining the effects of the intervention on feelings towards exercise and qualitative data from the interviews.

ELIGIBILITY:
Inclusion Criteria:

* lives in the US
* 18 years old or older
* desires to increase activity through structured exercise
* has an iPhone that can send/receive text messages and an Apple Watch

Exclusion Criteria:

* medically advised not to exercise

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 200 (Actual)
Dates: Start 2023-05-31 (Actual); Primary Completion 2023-11-01 (Actual); Study Completion 2023-11-30 (Actual)

PRIMARY OUTCOMES:
Calories burned in planned exercise session | 4 hours
  Calories burned during the four-hour time window when participants planned to exercise

SECONDARY OUTCOMES:
Change from Baseline Expected Post-exercise affect at 9 weeks | At study completion, 9 weeks after enrollment
  Participants will be asked question about their expected post-exercise affect at the beginning and end of the 9 week study
Change from Baseline in other affective attitude measures at 9 weeks | At study completion, 9 weeks after enrollment
  Participants will be asked additional questions about their affective attitudes towards and valuations of exercise at the beginning and end of the 9 week study

CONTACTS AND LOCATIONS:
Locations (1):
- University of Michigan, Ann Arbor, Michigan, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Mishra SR, Dempsey W, Klasnja P. A Text Messaging Intervention for Priming the Affective Rewards of Exercise in Adults: Protocol for a Microrandomized Trial. JMIR Res Protoc. 2023 Sep 1;12:e46560. doi: 10.2196/46560. PMID 37656493